CLINICAL TRIAL: NCT02716181
Title: A Double-Blind Randomized Placebo-Controlled Trial to Evaluate the Efficacy of the "Атопик Soothing Cream" in Children With Mild to Moderate Atopic Dermatitis
Brief Title: Efficacy of the "Атопик Soothing Cream" in Children With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avanta Trading Ltd. (Industry)
Collaborators: Samara State Medical University (Other); Prof. Zvulunov Alex, Pediatric Dermatology Clinic, Kfar-Saba, Israel. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 166-2015
Record Dates: First submitted 2016-03-13; First posted 2016-03-23 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2016-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Topical therapy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- "Атопик" phase 1 (Active Comparator): For the first phase of the study, subjects will be randomized to receive treatment with "Атопик Soothing Cream".
  Interventions: Device: "Атопик Soothing Cream"; Device: Placebo
- Placebo - phase 1 (Placebo Comparator): For the first phase of the study, subjects will be randomized to receive treatment with Placebo Cream.
  Interventions: Device: "Атопик Soothing Cream"; Device: Placebo
- "Атопик" phase 2 (Active Comparator): The second phase of the study is an open-label extension with all subjects receiving "Атопик Soothing Cream".
  Interventions: Device: "Атопик Soothing Cream"; Device: Placebo
- Placebo - phase 2 (Placebo Comparator): The second phase of the study is an open-label extension with all subjects receiving "Атопик Soothing Cream".
  Interventions: Device: "Атопик Soothing Cream"; Device: Placebo

INTERVENTIONS:
Device: "Атопик Soothing Cream" — Topical application of a study cream to involved skin areas twice a day.
Device: Placebo — Topical application of a study placebo cream to involved skin areas twice a day.

SUMMARY:
A Double-Blind Randomized Placebo-Controlled Trial to Evaluate the Efficacy of the "Атопик Soothing Cream" in Children with Mild to Moderate Atopic Dermatitis

DETAILED DESCRIPTION:
"Атопик Soothing Cream" is a lipid complex composed of barley grain, Butyrospermum Parkii and Argania Spinosa Kernel oil, in a mixture with panthenol and bisabolol.

Investigators concure that combination of these substances in "Атопик Soothing Cream" will be efficacious non-steroidal treatment of Atopic Dermatiti ( AD).

ELIGIBILITY:
Inclusion Criteria:

* Must have clinical diagnosis of mild to moderate atopic dermatitis (AD) at both Screening and Baseline Visits, defined as IGA score of 2 or 3 ( Rothe 1996) or EASI score between 2 and 21 (Leshem 2015)
* Must have AD affecting >5% total body surface area (TBSA) at Baseline
* History of AD for at least 3 months prior to Baseline
* Informed consent/assent in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guideline and applicable regulations, before completing any study-related procedures

Exclusion Criteria:

* Use of topical corticosteroids within 7 days prior to Baseline
* Use of systemic corticosteroids, topical calcineurin inhibitors, photo-therapy (PUVA, UVB) or immunosuppressive therapy (eg, cyclosporine) within 14 days prior to Baseline
* Subjects that require systemic therapy for the treatment of AD
* Use of systemic anti-infective or antibiotic treatment within 14 days prior to Baseline
* Subjects who present with clinical conditions other than AD that may interfere with the evaluation (eg, generalized erythroderma, acne, Netherton's Syndrome, psoriasis)
* Any clinically significant skin disease other than AD
* Secondary infection of AD (bacterial, viral or fungal) within the skin area under study or open skin infections in any area at Baseline
* History of severe anxiety and/or depression; any history of suicide attempt
* Subjects with a history of human immunodeficiency virus (HIV) as determined by medical history
* Subjects who, in the opinion of the Investigator(s), would be non-compliant with the visit schedule or study procedures
* Participation in any other investigational trial within 6 weeks of Baseline, or during study conduct
* Chronic condition(s) which are either unstable or not adequately controlled
* Drug or alcohol abuse, mental dysfunction, or other condition limiting the subject's ability to be compliant with study-related procedures
* Any medical condition that may, in the opinion of the Investigator(s), preclude the safe administration of test article or safe participation in the study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Investigators' Global Assessment score | 28 days

SECONDARY OUTCOMES:
Eczema Area & Severity Index (EASI) | 28 days
Pruritus intensity | 28 days
  Visual Analog Scale

OTHER OUTCOMES:
Trans-Epidermal Water Loss | 28 days
Stratum Corneum Capacitance | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alex Zvulunov, MD, Study Director — Prof. Alex Zvulunov, Pediatric Dermatology Clinic, Israel
Locations (1):
- Pediatric Allergy-Immunology, Department of Pediatrics, Institute of Professional Education, Samara, Russia

IPD SHARING:
Plan to Share IPD: Yes
Clinical parameters at the entry and at the end of study might be shared.

REFERENCES:
- [Background] Maurya AK, Singh M, Dubey V, Srivastava S, Luqman S, Bawankule DU. alpha-(-)-bisabolol reduces pro-inflammatory cytokine production and ameliorates skin inflammation. Curr Pharm Biotechnol. 2014;15(2):173-81. doi: 10.2174/1389201015666140528152946. PMID 24894548
- [Background] Ebner F, Heller A, Rippke F, Tausch I. Topical use of dexpanthenol in skin disorders. Am J Clin Dermatol. 2002;3(6):427-33. doi: 10.2165/00128071-200203060-00005. PMID 12113650
- [Result] Jirabundansuk P, Ophaswongse S, Udompataikul M. Comparative trial of moisturizer containing spent grain wax, Butyrospermum parkii extract, Argania spinosa kernel oil vs. 1% hydrocortisone cream in the treatment of childhood atopic dermatitis. J Med Assoc Thai. 2014 Aug;97(8):820-6. PMID 25345257